CLINICAL TRIAL: NCT05213117
Title: Optimizing Medical "Teaming" on Resident Based Teams
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Kathleen Finn, Senior Associate Program Director for Resident Development, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Protocol #: 2019P000534
Record Dates: First submitted 2021-12-13; First posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Inter-professional Relations
MeSH Terms: interventions — Nursing

STUDY DESIGN:
Intervention Model Description: The investigators plan to randomize 16-18 Post Graduate Year (PGY)-1 residents in internal medicine at Massachusetts General Hospital from the possible 74 PGY-1 incoming residents who agree to partake in the study to one general medicine clinical floor for the academic year. These co-localized residents will complete 16-20 weeks of scheduled rotation time on White 9. Similarly, the investigators plan to randomize 6-8 PGY-2 residents from a possible group of 64 PGY-2 residents who agree to participate in the study to one general medical clinical floor for the academic year. These participants will complete 4-6 weeks of scheduled rotation time on White 9. Rotations will be completed in the normal 2 or 4 week block rotations, randomly assigned throughout the academic year.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Co-localized Residents (Experimental): Investigators plan to randomize 15 PGY-1 residents in internal medicine from the possible 74 PGY-1 incoming residents who agree to partake in the study, to one general medicine clinical floor for the academic year. These co-localized residents will complete 16-20 weeks of scheduled rotation time on White 9
  Interventions: Behavioral: Co-Localization with Nursing
- Normally Schedule Residents (No Intervention): The control arm will consist of 18 PGY-1 residents who are scheduled by the residency program's algorithm in the usual fashion to complete general medicine rotations on 5 difference clinical floors. The 18 active comparator participants will be selected based on completing one of four general medicine rotation on the control floor White 8. These participants will then be followed while completing the remaining general medicine rotations on all clinical floors.

INTERVENTIONS:
Behavioral: Co-Localization with Nursing — Co-localize 15 residents to one of 6 general medical floors to complete all 8 weeks of general medicine on this floor
  Arms: Co-localized Residents

SUMMARY:
The main objective of this study is to evaluate the colocalization of internal medicine residents on one clinical inpatient hospital floor for all general medicine block rotations during the 2019-2020 academic year. Specifically, the aims of the study are to determine if co-localization improves familiarity with nursing staff, which in turn, improves team work, psychological safety, patient care and reduces burnout. The investigators' hypothesis is that co-localization will increase familiarity between residents and nurses and result in improved psychological safety, team work and patient outcomes.

DETAILED DESCRIPTION:
Teamwork is critical in delivering high quality medical care. Failures in team communication and coordination have been cited as significant contributors to medical errors. In large teaching hospitals, patients receive care from transiently formed teams of nurses and residents who may only work together for as little as two weeks, as residents rotate through many clinical floors due to the complexity of resident scheduling. Unlike more established teams that work together over long periods of time, these transient groups are called "teaming;" a process where a group of diverse providers, with different roles, outlooks and levels of professional training transiently come together to carry out complex tasks. (Reference: Dr. Amy Edmondson, Harvard Business School) A key risk in "teaming" is the lack of familiarity of team members as studies suggest familiarity promotes an environment of psychological safety, where team members feel safe speaking up, asking for help and admitting errors. These skills are important for both team work and patient safety. The investigators hypothesize that in large residency programs where resident rotate on multiple floors, it is possible to improve the quality of "teaming" by increasing the frequency with which smaller groups of residents and nurses work together. As a result, the investigators propose a randomized controlled trial on an inpatient general medical floor to study the effect of co-localizing residents with nursing staff. One cohort of residents will be assigned to complete all general medical rotations on a single floor for the academic year. The investigators will assess the impact on psychological safety, team work and patient care. The investigators hypothesize by co-localizing residents with nursing, while these "teaming" are still transient, the slight increase in familiarity will promote a culture of psychological safety and improve team work. If benefits are found, resident scheduling can be adjusted in subsequent years.

ELIGIBILITY:
Inclusion Criteria:

* All incoming PGY-1 residents who volunteer to be randomized

Exclusion Criteria:

* Any incoming PGY-1 resident who declines to be randomized

Min Age: 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2020-06-24 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
Teamwork assessed by Simulation about Shortness of Breath | This simulation will be conducted at 6 months in this 12month study
  Simulation of an inpatient clinical scenario will be conducted. This simulation about shortness of breath will be run with teams consisting of two residents and two nurses. These interdisciplinary teams will be asked to manage a patient together. All residents and nurses in the study will be asked to participate in the simulation. The simulations will be recorded. Blinded reviewers will view these simulations later and will score the team's performance using an published Oxford NOTECH simulation teamwork assessment tool. The assessment tool is designed to identify higher functioning teams by evaluating leadership, communication, shared mental models and utilization of resources.
Teamwork assessed by Simulation about Negotiation with Angry Patient | This simulation will be conducted at 12 months in this 12month study
  Simulation of an inpatient clinical scenario will be conducted. This simulation about negotiating with an angry patient will be run with teams consisting of two residents and two nurses. These interdisciplinary teams will be asked to manage a patient together. All residents and nurses in the study will be asked to participate in the simulation. The simulations will be recorded. Blinded reviewers will view these simulations later and will score the team's performance using an published Oxford NOTECH simulation teamwork assessment tool. The assessment tool is designed to identify higher functioning teams by evaluating leadership, communication, shared mental models and utilization of resources.

SECONDARY OUTCOMES:
Psychological Safety | Residents and Nurses will be surveyed at 6 months in this 12 month study
  A survey tool has been developed for both residents and nurses. The survey tool asks questions using a 5 point Likert scale about psychological safety, communication and teamwork. The questions were modified based on prior published work by Dr. Amy Edmondson at the Harvard Business School. The survey will be used to evaluate the residents and nurses perception of teamwork and psychological safety.
Psychological Safety | Residents and Nurses will be surveyed at 12 months in this 12 month study
  A survey tool has been developed for both residents and nurses. The survey tool asks questions using a 5 point Likert scale about psychological safety, communication and teamwork. The questions were modified based on prior published work by Dr. Amy Edmondson at the Harvard Business School. The survey will be used to evaluate the residents and nurses perception of teamwork and psychological safety.
Communication between Nurses and Interns | Observation will start at 6 months in this 12 month study and continue through study completion, an average of 6 months
  A time motion study will be conducted where an observer with an Apple iPad will observe rounds with nurses and interns. The observer will record the amount of time each individual is speaking, the length of rounds and the number of patients rounded on.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen F Finn, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and results
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be published in 2022
Access Criteria: Plan to publish in 2022

REFERENCES:
- [Derived] Iyasere CA, Wing J, Martel JN, Healy MG, Park YS, Finn KM. Effect of Increased Interprofessional Familiarity on Team Performance, Communication, and Psychological Safety on Inpatient Medical Teams: A Randomized Clinical Trial. JAMA Intern Med. 2022 Nov 1;182(11):1190-1198. doi: 10.1001/jamainternmed.2022.4373. PMID 36215043